CLINICAL TRIAL: NCT06283797
Title: Assessment of the Efficacy of Automated Insulin Therapy (Artificial Pancreas) Early Initiated After Diagnosis on Blood Glucose Control in Children and Adolescents With Type 1 Diabetes: Randomized Comparison With Conventional Insulin Therapy on 1 Year, Followed by an Optional Extension on 1 Year
Brief Title: Efficacy of Automated Insulin Therapy Early Initiated After Diagnosis on Blood Glucose Control in Children and Adolescents With Type 1 Diabetes
Acronym: APATDIAGNOSIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Hopital Universitaire Robert-Debre (Other); University Hospital, Tours (Other); University Hospital, Angers (Other Government); University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL22_0346; 2023-A01661-44 (Other: ANSM)
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Diabetes
Keywords: Type 1 diabetes; Children and adolescents; Recent diagnosis of diabetes; Automated insulin delivery; Randomized control
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Randomized control study in parallel groups, followed by a non randomized extension
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Automated insulin delivery (Experimental): Participants will use an automated insulin delivery system with study CGM
  Interventions: Device: OmniPod 5; Device: Dexcom G6; Other: PAID questionnaires
- Conventional insulin therapy (Active Comparator): Participants will use multiple insulin daily insulin injections or insulin pump with study CGM
  Interventions: Device: Dexcom G6; Other: PAID questionnaires

INTERVENTIONS:
Device: OmniPod 5 — Participants will be trained to use OmniPod 5 to treat type 1 diabetes for 1 year
  Arms: Automated insulin delivery
Device: Dexcom G6 — Participants will use Dexcom G6 for continuous glucose monitoring
Other: PAID questionnaires — At visits 3, 7 and 11, parents/guardians and patients aged between 8 and 17 will complete diabetes-related problem questionnaires (PAID-PR, PAID-Peds)

SUMMARY:
The main objective is to assess whether hybrid closed-loop (HCL) insulin delivery initiated early after diagnosis of Type 1 diabetes (T1D) allows a better efficacy on glucose control than conventional standard insulin therapy with multiple daily insulin injections (MDI) or insulin pumps after one year of use.

The secondary objectives are to assess whether HCL initiated early after diagnosis of T1D allows: (1) Higher time spent with glucose level in the near-normal range, (2) Lower time spent in hypoglycemia and hyperglycemia, (3) Lower glucose variability, (4) Lower perceived burden of diabetes management, (5) Better preserved endogenous insulin secretion, all the above after one year of use, (6) Lower occurrence of interventions for hypoglycemia, versus conventional standard insulin therapy with MDI or insulin pump.

An optional 1-year extension aims at assessing: (1) Sustainability of above mentioned parameters over a second year of HCL use in the group who started HCL early after diagnosis, (2) Efficacy on glucose control according to the above mentioned parameters when HCL is initiated early after diagnosis vs. after 1 year in the control group of the randomized phase.

DETAILED DESCRIPTION:
This is a prospective, open-label, multicenter, 1-year randomized control trial, followed by an optional 1-year extension. Based upon computed number of needed participants, 112 patients aged 2-17.9 with a diagnosis of T1D within 3-6 months, trained for meal carbohydrate counting (independently or with their parents/guardians) will be enrolled after written informed consent. All participants will be trained to guide their insulin doses from the data of Dexcom G6 CGM system during a 30-day run-in phase. Downloaded CGM data, measured HbA1c and stimulated C-peptide levels and answered study questionnaires at randomization visit will serve as baseline reference. The participants will be randomized 1:1 to either HCL or their usual insulin therapy by MDI or insulin pump (control group). Participants allocated to HCL and their parents/guardians will be trained to the study AID system. Safety phone visits will be scheduled 48 hours, 1 week and 2 weeks after HCL initiation. The participants randomized to the control group will go on using their usual insulin treatment while using the Dexcom G6 data to guide their insulin doses. Outpatient visits will occur every 3 months for one year in both study groups for the monitoring of glucose control (and HCL system functioning if applicable), safety and protocol adherence. At one year, study primary endpoint will be assessed, as well as all secondary study endpoints using a repeated measure ANOVA with within/between factor. After one year, the participants and their parents/guardians of the control group will be offered to switch to HCL with the study system for one year while the initial HCL system group will be offered to keep this therapy for an additional year, with quarterly monitoring visits in the whole population for this optional extension phase of the study. At the end of this extension, all study endpoints will be re-assessed.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 2 and 17.9 years
* Diagnosis of type 1 diabetes since at least 3 months and up to 6 months based upon WHO criteria
* Identification of at least one positive plasma auto-antibody among anti-GAD, anti-IA2, anti-ZnT8 and anti-insulin
* Treatment by multiple-daily insulin injections or insulin pump. An insulin pump with a function of stopping the pump in case of predicted hypoglycaemia is allowed.
* Patient and/or parents/guardians trained in carbohydrate counting
* Patient and/or parents/guardians must have a smartphone that supports the Dexcom G6 app download and participants must be willing to use Dexcom G6 sensor and app throughout the study

Exclusion Criteria:

* Unwillingness of one parent or the legally responsible party to participate in insulin treatment
* Any associated chronic disease or therapy (except insulin or L thyroxin at stable dose) affecting glucose metabolism
* Therapy by automated insulin delivery using an insulin pump connected to continuous glucose monitoring sensor with a control algorithm (hybrid closed-loop system)
* Cutaneous allergy or contact dermatitis to device (CGM or pod) adhesives
* Insufficient vision and/or hearing to recognise all the functions of the Omnipod 5 system, including alerts, alarms and reminders in accordance with the instructions of utilization
* Impaired cognitive or psychological abilities of the patient and/or his/her parents or the legally responsible party which may result in defective adherence to study procedures
* Active enrolment in another clinical trial or administration of an unapproved drug within the last 4 weeks before the screening date
* Subject who is in a dependency or employment with the sponsor or the investigator
* No signed informed consent form by the patient and his/her parents/legally responsible party
* Subjects unable to attend all scheduled visits and to comply with all trial procedures
* Law protected or deprived of liberty subject
* Pregnant and breastfeeding women
* Subjects no covered by public health insurance

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-06-29 (Estimated); Study Completion 2027-06-29 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c) level | At 1 year follow-up
  Change in the HbA1c level, measured by HPLC method, from the start of the randomized study phase to the end of this 1-year study phase

SECONDARY OUTCOMES:
Percent of time spent in the 70-180 mg/dl glucose range | At 1 year follow-up
  Continuous glucose monitoring
Percent of time spent in the 70-140 mg/dl glucose range | At 1 year follow-up
  Continuous glucose monitoring
Mean glucose level | At 1 year follow-up
  Continuous glucose monitoring
Percent of time spent with glucose level below 70 mg/dl | At 1 year follow-up
  Continuous glucose monitoring
Percent of time spent with glucose level below 54 mg/dl | At 1 year follow-up
  Continuous glucose monitoring
Percent of time spent with glucose level above 180 mg/dl | At 1 year follow-up
  Continuous glucose monitoring
Percent of time spent with glucose level above 250 mg/dl | At 1 year follow-up
  Continuous glucose monitoring
Coefficient of glucose variability | At 1 year follow-up
  Continuous glucose monitoring
Score of PAID questionnaire for parents | At 1 year follow-up
  Change of score of PAID-PR in order to assess perceived burden of diabetes management
Score of PAID questionnaire for children | At 1 year follow-up
  Change of score of PAID-Peds (age: 8-17) in order to assess perceived burden of diabetes management
Stimulated plasma C-peptide level 10-min after 1mg IV glucagon | At 1 year follow-up
  Changes in stimulated plasma C-peptide level 10-min after 1mg IV glucagon in order to assess preserved endogenous insulin secretion
Number of needed interventions by the parents/guardians or care providers | At 1 year follow-up
  Number of needed interventions by the parents/guardians or care providers to treat hypoglycemia, between randomized groups in order to assess occurrence of interventions for hypoglycemia

OTHER OUTCOMES:
Change of HbA1c level between 1st and 2nd year of use in the group who started HCL early after diagnosis | At 2 years follow-up
Change of percent of time spent in the 70-180 mg/dl glucose range between 1st and 2nd year of use in the group who started HCL early after diagnosis | At 2 years follow-up
Change of percent of time spent in the 70-140 mg/dl glucose range between 1st and 2nd year of use in the group who started HCL early after diagnosis | At 2 years follow-up
Change of mean glucose level between 1st and 2nd year of use in the group who started HCL early after diagnosis | At 2 years follow-up
Change of percent of time spent with glucose level below 70 mg/dl between 1st and 2nd year of use in the group who started HCL early after diagnosis | At 2 years follow-up
Change of percent of time spent with glucose level below 54 mg/dl between 1st and 2nd year of use in the group who started HCL early after diagnosis | At 2 years follow-up
Change of percent of time spent with glucose level above 180 mg/dl between 1st and 2nd year of use in the group who started HCL early after diagnosis | At 2 years follow-up
Change of percent of time spent with glucose level above 250 mg/dl between 1st and 2nd year of use in the group who started HCL early after diagnosis | At 2 years follow-up
Change of coefficient of glucose variability between 1st and 2nd year of use in the group who started HCL early after diagnosis | At 2 years follow-up
Change of score of PAID questionnaire for parents between 1st and 2nd year of use in the group who started HCL early after diagnosis | At 2 years follow-up
Change of score of PAID questionnaire for children between 1st and 2nd year of use in the group who started HCL early after diagnosis | At 2 years follow-up
Change of stimulated plasma C-peptide level 10-min after 1mg IV glucagon between 1st and 2nd year of use in the group who started HCL early after diagnosis | At 2 years follow-up
Change of number of needed interventions by the parents/guardians or care providers between 1st and 2nd year of use in the group who started HCL early after diagnosis | At 2 years follow-up
Difference in the HbA1c level between the 2 initially randomized groups at the end of the extension period | At 2 years follow-up
Difference in the percent of time spent in the 70-180 mg/dl glucose range between the 2 initially randomized groups at the end of the extension period | At 2 years follow-up
Difference in the percent of time spent in the 70-140 mg/dl glucose range between the 2 initially randomized groups at the end of the extension period | At 2 years follow-up
Difference in the mean glucose level between the 2 initially randomized groups at the end of the extension period | At 2 years follow-up
Difference in the percent of time spent with glucose level below 70 mg/dl between the 2 initially randomized groups at the end of the extension period | At 2 years follow-up
Difference in the percent of time spent with glucose level below 54 mg/dl between the 2 initially randomized groups at the end of the extension period | At 2 years follow-up
Difference in the percent of time spent with glucose level above 180 mg/dl between the 2 initially randomized groups at the end of the extension period | At 2 years follow-up
Difference in the percent of time spent with glucose level above 250 mg/dl between the 2 initially randomized groups at the end of the extension period | At 2 years follow-up
Difference in the coefficient of glucose variability between the 2 initially randomized groups at the end of the extension period | At 2 years follow-up
Difference in the score of PAID questionnaire for parents between the 2 initially randomized groups at the end of the extension period | At 2 years follow-up
Difference in the score of PAID questionnaire for children between the 2 initially randomized groups at the end of the extension period | At 2 years follow-up
Difference in the stimulated plasma C-peptide level 10-min after 1mg IV glucagon between the 2 initially randomized groups at the end of the extension period | At 2 years follow-up
Difference in the number of needed interventions by the parents/guardians or care providers between the 2 initially randomized groups at the end of the extension period | At 2 years follow-up
Incidence of treatment-emergent SUSARs, SAEs, ARs and AEs | At 2 years follow-up
  Evaluated at each visit until the end of study in order to assess the safety of studied intervention
Relatedness of treatment-emergent SUSARs, SAEs, ARs and AEs | At 2 years follow-up
  Evaluated at each visit until the end of study in order to assess the safety of studied intervention
Severity of treatment-emergent SUSARs, SAEs, ARs and AEs | At 2 years follow-up
  Evaluated at each visit until the end of study in order to assess the safety of studied intervention

CONTACTS AND LOCATIONS:
Overall Officials: Eric RENARD, MD, Principal Investigator — University Hospital, Montpellier
Locations (4):
- France (4):
  - University Hospital, Angers, Angers
  - University Hospital, Montpellier, Montpellier
  - Robert Debré Hospital, AP-HP, Paris
  - University Hospital, Tours, Tours